CLINICAL TRIAL: NCT05623579
Title: Effect of Therapeutic Education on Pain Intensity and BDNF Levels in Patients With Chronic Pain
Brief Title: Education on BDNF on Pain Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022A36005
Record Dates: First submitted 2022-10-25; First posted 2022-11-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: BDNF; Pain Neuroscience Education; Exercise
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pain Education plus Exercise
  Interventions: Behavioral: Pain Neuroscience Education; Behavioral: Exercise
- Control (Active Comparator): Exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — 8 Sessions of different pain education interventions
  Arms: Intervention
Behavioral: Exercise — 12 Sessions of Aerobic Exercise

SUMMARY:
The promotion of neuroplasticity in conjunction with strategies for restructuring maladaptive cognitions that largely cause the activation of neural networks that contribute to the perpetuation of pain is therefore a fundamental neurophysiological principle for establishing a neurophysiological basis for pain.

perpetuation of pain, is therefore a fundamental neurophysiological principle for establishing physiotherapy therapeutic to establish therapeutic strategies from physiotherapy that contribute to improve the quality of life of patients with chronic pain. patients with chronic pain.

Based on the theory that neurotrophic factors such as BDNF play a fundamental role in the initiation and or maintenance of hyperexcitability of central neurons in pain, we consider that the levels of this neurotrophic factor, such as BDNF, may have an important role in the perpetuation of pain.

that the levels of this neurotrophic factor may be modified by the application of a therapeutic education protocol, favoring therapeutic education protocol, favoring a reduction in pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18 to 65 years with musculoskeletal pain for a minimum of 3 months
* patients recruited by information pamphlets from the university clinic of the Rey Juan Carlos University, and CSEU La Salle
* not having received physiotherapy treatment for this same process in the last 3 months.
* ability to perform all the clinical tests and to understand the study process, as well as to obtain informed consent.

Exclusion Criteria:

- Systemic, neurological, oncological or inflammatory diseases; psychiatric pathologies, pregnancy, type II diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 36 weeks
  Pain intensity assessed with the 100 mm Visual Analog Scale, in which the patient is asked about his or her pain level at that moment, with one side being "no pain" and the other extreme being "the worst pain imaginable".

SECONDARY OUTCOMES:
BDNF level | 36 weeks
  BDNF level measured in blood serum by ELISA kit at baseline and at the end of the intervention.
Anxiety and Depression (HADS) | 36 weeks
  Anxiety and depression will be assessed using the Spanish validated version of the HADS. The HADS is a self-administered measure with 14 items in total that ask the client to reflect on their mood in the past week. Seven items assess depression, 5 of which are markers for anhedonia (an inability to experience pleasure), and 2 concern appearance and feelings of slowing down. Seven items assess anxiety, of which 2 assess autonomic anxiety (panic and butterflies in the stomach), and the remaining 5 assess tension and restlessness (Dunbar, Ford, Hunt, & Der, 2000).
Quality of life (EQ-5D) | 36 weeks
  The EQ-5D is a generic HRQoL. HRQoL that can be used both in relatively healthy individuals (general population) and in groups of patients with different pathologies. The individual assesses his or her own health status, first in levels of severity by dimensions and then on a more general visual analog scale (VAS).The third element of the EQ-5D is the index of social values that is obtained for each health state generated by the instrument. In this part of the questionnaire, the individual must mark the level of severity corresponding to his or her health status in each of the dimensions health status in each of the dimensions, referring to the same day on which the same day the questionnaire is completed.
Pain Catastrophism (PCS) | 36 weeks
  Pain Catastrophism will be measured with the Spanish version of the Pain Catastrophism Scale. The Pain Catastrophizing Scale (PCS) is a 13-item self-report questionnaire considered to be the most frequent and extensively studied tool to assess pain catastrophizing for chronic pain. Good levels of content and construct validity, internal consistency and test-retest reliability of the PCS have been reported in studies examining different musculoskeletal disorders and different language versions.
Pain Severity Level (GCPS-R) | 36 weeks
  Pain severity will be measured Chronic Pain Grading Scale Description: A measure of pain intensity and interference with normal daily activities.
  Format: 7 items
  Scoring: Scores for 6 of the items range from 0 (no pain) to 10 (pain as bad as it could be). The one remaining item requires filling in the number of days that pain has kept respondents from their typical activities.
  Scores classify respondents into one of 4 levels of pain intensity and activity interference:
  Low disability and low pain intensity Low disability and high pain intensity High disability and moderate limitation of activities High disability and severe limitation of activities
Oxygen Saturation (SpO2) | 36 weeks
  measured with a finger pulse oximeter: A normal ABG oxygen level for healthy lungs falls between 80 and 100 millimeters of mercury (mm Hg).
Heart rate (HR) | 36 weeks
  measured with a finger pulse oximeter: A normal Heart Rate is between 60 and 120 pulse per minute.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clínica URJC, Alcorcón, Madrid
  - IRF La Salle, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Result] Andias R, Neto M, Silva AG. The effects of pain neuroscience education and exercise on pain, muscle endurance, catastrophizing and anxiety in adolescents with chronic idiopathic neck pain: a school-based pilot, randomized and controlled study. Physiother Theory Pract. 2018 Sep;34(9):682-691. doi: 10.1080/09593985.2018.1423590. Epub 2018 Jan 10. PMID 29319386